CLINICAL TRIAL: NCT04971941
Title: Evaluation of the Dental Vibe Injection Comfort System
Acronym: DVRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, jeffry_shaefer@hms.harvard.edu, Assistant Professor of Oral and Maxillofacial Surgery, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB14-2778
Record Dates: First submitted 2021-02-28; First posted 2021-07-22 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia, Local; Pain
Keywords: Anesthesia, local; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- DV3 with first LB injection (Active Comparator): Use of Dental Vibe with first long buccal block
  Interventions: Device: Dental Vibe
- DV3 with first LB and with IAN (Active Comparator): Dental Vibe with first long buccal injection and inferior alveolar block
  Interventions: Device: Dental Vibe
- DV3 with 2nd LB (Experimental): Use of DentalVibe with 2nd Long Buccal injection
  Interventions: Device: Dental Vibe
- DV3 with 2nd LB and IAN (Experimental): Use of DentalVibe with 2nd long buccal and inferior alveolar nerve block
  Interventions: Device: Dental Vibe

INTERVENTIONS:
Device: Dental Vibe — Use of Dental Vibe during dental anesthesia intervention

SUMMARY:
This study investigated the Dental Vibe Injection Comfort System (DV), developed to lessen anesthesia pain through pulsed vibration, a form of counter-stimulation. The study's aims were to evaluate DV's efficacy in reducing pain/discomfort from intra-oral long buccal (LB) and inferior alveolar nerve (IAN) injections and the time needed to achieve complete anesthesia during an IAN block.

DETAILED DESCRIPTION:
Objective: Pain from local anesthesia injections can be reduced by distraction and counter-stimulation techniques. This study investigated the Dental Vibe Injection Comfort System (DV), developed to lessen anesthesia pain through pulsed vibration, a form of counter-stimulation.

Design: Our study's aims were to evaluate DV's efficacy in reducing pain/discomfort from intra-oral long buccal (LB) and inferior alveolar nerve (IAN) injections and the time needed to achieve complete anesthesia during an IAN block.

Methods: The sixty subjects, equally split by sex, ages 21-32, rated injection pain on a visual analog scale and discomfort, unpleasantness, and difficulty in enduring the injection on a modified symptom severity index. Each subject received bilateral LB injections and an IAN block. Using block design, DV Generation 3 (DV3) was randomly assigned to either the first or second LB injection and to thirty subjects on their third injection, the IAN block. No topical anesthesia was applied.

ELIGIBILITY:
Inclusion Criteria: Able to volunteer for dental anesthesia -

Exclusion Criteria: Non volunteer

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffry R Shaefer, DDS MS MPH, Principal Investigator — Harvard School of Dental Medicine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 subjects participated in this study. Each participant had 3 procedures done (bilateral buccal nerve blocks one with or without the use of Dentalvibe, and then one inferior alveolar nerve (IAN) block for which 30 subjects had it done with the Dentalvibe and 30 subjects had it done without the use of the Dentalvibe. The IAN blocks with or w/o the Dentalvibe was chosen randomly.and which side went first with or without the Dentalvibe was also chosen randomly.
Groups:
- DV3 With 1st LB Injection: This group had DV3 only with 1st Long Buccal injection
- DV3 With 1st LB Injection and IAN Block (3rd Injection): This group had DV3 with their first Long Buccal injection and their IAN block injection
- DV3 With 2nd LB Injection: This group had the DV3 used only during their 2nd long buccal injection
- DV3 With 2nd LB Injection and IAN Block (3rd Injection): This group had the DV3 used with their 2nd Long Buccal injection and during their IAN injection
Period: Overall Study
Arm/Group | DV3 With 1st LB Injection | DV3 With 1st LB Injection and IAN Block (3rd Injection) | DV3 With 2nd LB Injection | DV3 With 2nd LB Injection and IAN Block (3rd Injection)
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 60 subjects participated in the study. In the long bucal portion each subject had an injection with and without the Dental Vibe with the DV3 being used first on the left side in 30 subjects and first on the right side in 30 subjects while in the IAN part of the study 30 had an injection without the Dentalvibe and 30 with the Dentalvibe. Pain and tolerability, and time to complete anesthesia were compared.
Groups:
- DV3 With 1st LB Injection: DV3 with First Long Buccal Use of Dental Vibe during dental anesthesia intervention
- DV3 With 1st LB Injection and IAN Block (3rd Injection): Dental Vibe with first long buccal injection and IAN
  Dental Vibe: Use of Dental Vibe during dental anesthesia intervention
- DV3 With 2nd LB Injection: DV3 with 2nd Long Buccal Injection
  Dental Vibe: Use of Dental Vibe during dental anesthesia intervention
- DV3 With 2nd LB Injection and DV3 With 2nd LB and IAN Injections: DV3 with 2nd Long Buccal Injection and also with Inferior Alveolar injection
- Total: Total of all reporting groups
Arm/Group | DV3 With 1st LB Injection | DV3 With 1st LB Injection and IAN Block (3rd Injection) | DV3 With 2nd LB Injection | DV3 With 2nd LB Injection and DV3 With 2nd LB and IAN Injections | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 15 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (1.5) | 24 (1) | 27 (1.5) | 26 (1) | 25 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 8 | 7 | 30
  Male | 8 | 7 | 7 | 8 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 15 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: VAS
Description: VAS (visual analog scale) measured pain during anesthesia procedure on a scale from 0-10 with 0 being no pain and 10 being the most intense pain. The lowest number is the best outcome.
Time Frame: Measured during anesthesia procedure by the subject and recorded after each individual anesthesia procedure, an average of one minute
Population: Subjects getting IAN with or without DV, LB with DV used first, LB with DV used second
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Inferior Alveolar Block: Use of DentalVibe with or without inferior alveolar nerve block
  Use of DentalVibe during dental anesthesia intervention compared to inferior alveolar nerve block without DentalVibe
- LB Injection With DV First: Each subject had bilateral LB injections. These subjects had use of Dental Vibe during dental anesthesia intervention for the initial LB injection as compared to the second LB done on opposite side w/o DV
- Long Buccal Injection With DV Second: Dental Vibe: Use of Dental Vibe during dental anesthesia intervention after LB w/o DentalVibe was done initially with opposite side then receiving a LB with DentalVibe
Arm/Group | Inferior Alveolar Block | LB Injection With DV First | Long Buccal Injection With DV Second
Number analyzed (Participants) | 60 | 30 | 30
score on a scale
  with dental vibe: number analyzed (Participants) | 30 | 30 | 30
  with dental vibe | 2.5 (1.48) | 2.3 (1.21) | 2.7 (1.46)
  without dental vibe: number analyzed (Participants) | 30 | 30 | 30
  without dental vibe | 4.2 (2.17) | 3.3 (1.75) | 4.0 (1.74)
Statistical Analysis 1: Comparison: Inferior Alveolar Block; Sample size estimation from Nanitsos 2010: Using the P value from the paired T test with 61 degrees of freedom the T statistic calculated at 4.365. From mean difference 9.3 SD was calculated as 16.66 for an effect size of 0.558. This generated a sample size of 44 subjects, receiving 2 injections (1 with DV3 and 1 without), is necessary to attain 95% power for a paired t-test comparing the 2 pain measures at a two-tailed alpha level of 0.05. P value for IAN; Test type: Superiority; p = 0.001, t-test, 2 sided — This P value applies to comparison of IAN with and without DentalVibe; df =58; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [0.4 to 2.1], Standard Deviation 2.17
Statistical Analysis 2: Comparison: LB Injection With DV First; Test type: Superiority; p = 0.02, t-test, 2 sided; df= 58; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-1.7 to -1.5], Standard Deviation 1.75
Statistical Analysis 3: Comparison: Long Buccal Injection With DV Second; Test type: Superiority; p = 0.004, t-test, 2 sided; Mean Difference (Net) = 1.2, 95% CI 2-sided [0.4 to 2.1], Standard Deviation 1.74

2. Secondary Outcome: SSI
Description: SSI measured tolerability, intensity, and unpleasantness of anesthesia procedure. Each has a scale from 0-28; with 0 being the least discomfort, least intolerable, and lowest intensity; whereas 28 is the most discomfort, most intolerable, and most intense.
Time Frame: measured by subject during procedure but recorded directly after each procedure
Population: scale from 0-28 with zero being non discomfort, completely tolerable, no unpleasantness
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SSI Tolerability Inf Alveolar Nerve Block: tolerability of injection rated on a scale from 0-28.
- SSI Discomfort Inf Alveolar Nerve Block: Intensity With and without use of dentalvibe scale 0-28
- SSI Unpleasantness IAN Block: with and without use of the Dentalvibe measured on a scale from 0-28
- SSI Tolerability LB Block DV First; SSI Discomfort LB DV First; SSI Unpleasantness LB With DV First: Long buccal (LB) nerve block with DV used first while opposite side LB done without DV done second
- SSI Tolerabilty Long Buccal Block DV Second: This group had LB without DV first and then DV was used for the opposite side LB injection
- SSI Discomfort LB DV Second: Long buccal (LB) nerve block without DV done first while opposite side LB with DV done second
- SSI Unpleasantness LB DV Second: Long buccal (LB) nerve block without DV done first while opposite side LB done with DV done second
Arm/Group | SSI Tolerability Inf Alveolar Nerve Block | SSI Discomfort Inf Alveolar Nerve Block | SSI Unpleasantness IAN Block | SSI Tolerability LB Block DV First | SSI Tolerabilty Long Buccal Block DV Second | SSI Discomfort LB DV First | SSI Discomfort LB DV Second | SSI Unpleasantness LB With DV First | SSI Unpleasantness LB DV Second
Number analyzed (Participants) | 60 | 60 | 60 | 30 | 30 | 30 | 30 | 30 | 30
score on a scale
  with dental vibe: number analyzed (Participants) | 30 | 30 | 30 | 30 | 30 | 30 | 30 | 30 | 30
  with dental vibe | 4.8 (3.02) | 6.2 (4.31) | 5.8 (4.04) | 4.0 (3.23) | 5.0 (3.77) | 5.3 (3.04) | 6.8 (4.5) | 5.3 (3.51) | 6.5 (4.36)
  without dental vibe: number analyzed (Participants) | 30 | 30 | 30 | 30 | 30 | 30 | 30 | 30 | 30
  without dental vibe | 8.9 (5.67) | 10.2 (5.42) | 9.8 (5.90) | 6.0 (4.66) | 7.6 (4.72) | 7.9 (4.21) | 9.1 (4.06) | 7.6 (4.67) | 8.8 (4.60)
Statistical Analysis 1: Comparison: SSI Tolerability Inf Alveolar Nerve Block; Test type: Superiority; p = 0.001, t-test, 2 sided — This P value applies to comparing IAN with or with DV as measured by SSI tolerability/ability to endure; Mean Difference (Net) = 4, 14% CI 2-sided [0.4 to 4.8]
Statistical Analysis 2: Comparison: SSI Discomfort Inf Alveolar Nerve Block; Test type: Superiority; p = 0.003, t-test, 2 sided
Statistical Analysis 3: Comparison: SSI Unpleasantness IAN Block; Test type: Superiority; p = 0.003, t-test, 2 sided
Statistical Analysis 4: Comparison: SSI Tolerability LB Block DV First; Test type: Superiority; p = 0.058, t-test, 2 sided
Statistical Analysis 5: Comparison: SSI Discomfort LB DV First; Test type: Superiority; p = 0.008, t-test, 2 sided
Statistical Analysis 6: Comparison: SSI Unpleasantness LB With DV First; Test type: Superiority; p = 0.044, t-test, 2 sided
Statistical Analysis 7: Comparison: SSI Tolerabilty Long Buccal Block DV Second; Test type: Superiority; p = 0.023, t-test, 2 sided
Statistical Analysis 8: Comparison: SSI Discomfort LB DV Second; Test type: Superiority; p = 0.042, t-test, 2 sided
Statistical Analysis 9: Comparison: SSI Unpleasantness LB DV Second; Test type: Superiority; p = 0.053, t-test, 2 sided

3. Secondary Outcome: Time in Minutes
Description: Time for complete inferior alveolar nerve block anesthesia with or without use of Dental Vibe measured in minutes. The time was recorded in minutes from when the anesthesia procedure was completed until the subject had a numb lip and could no longer feel cold (ice) applied to their ipsilateral canine tooth
Time Frame: After procedure until lip numbness, an average of four minutes
Population: time to complete mandibular anesthesia was measured
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Time for Complete Anesthesia for Inferior Alveolar Nerve Block: 30 participants for IAN complete block with and 30 without use of Dental Vibe
Arm/Group | Time for Complete Anesthesia for Inferior Alveolar Nerve Block
Number analyzed (Participants) | 60
minutes
  with Dentalvibe: number analyzed (Participants) | 30
  with Dentalvibe | 6 (5.0)
  without DentalVibe: number analyzed (Participants) | 30
  without DentalVibe | 7.8 (5.6)
Statistical Analysis 1: Comparison: Time for Complete Anesthesia for Inferior Alveolar Nerve Block; The null hypothesis is that there is no relation between use of DV and numb times. There were no studies from which to perform a power calculation for this outcome measure; Test type: Superiority; p = 0.459, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: During time of injection and until full anesthesia was achieved and during the post anesthesia period of 2 hours. The timeframe for adverse events was 2 hours.
Description: Common dental anesthesia procedures were done during this study with no serious side affects anticipated. No participants had mild or serious affects during his/her procedure
Groups:
- DV3 With First LB Block: Dental Vibe: Use of Dental Vibe during dental anesthesia intervention for Long Buccal only
- DV3 With 1st LB and IAN Block: Dental Vibe with long buccal injection and IAN block
- DV3 With 2nd LB: Dental Vibe: Use of Dental Vibe during dental anesthesia intervention for LB only
- DV3 With 2nd LB and IAN Block: Use of DV3 with LB and IAN blocks
- Inferior Alveolar Block: IAN block without DV
- LB Done First; LB Done 2nd: LB done without DV
Arm/Group | DV3 With First LB Block | DV3 With 1st LB and IAN Block | DV3 With 2nd LB | DV3 With 2nd LB and IAN Block | Inferior Alveolar Block | LB Done First | LB Done 2nd
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/60 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/60 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/60 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No